CLINICAL TRIAL: NCT04196881
Title: Effect of Attention Deficit Hyperactivity Disorder Knowledge Improvement Program on Male Primary School Teachers in Abha City: A Randomized Controlled Trial
Brief Title: Effect of Attention Deficit Hyperactivity Disorder Knowledge Improvement Program on Male Primary School Teachers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Abdullah Mohammed Alshehri, Principal Investigator, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADHD
Record Dates: First submitted 2019-12-08; First posted 2019-12-12 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: ADHD; Mental Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Saudi; Abha; Training; ADHD; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): group will receive training about ADHD
  Interventions: Other: Knowledge Improvement Program about ADHD
- Control (No Intervention): group will not receive training about ADHD

INTERVENTIONS:
Other: Knowledge Improvement Program about ADHD — This training program will cover an overview of ADHD, prevalence, causes, symptoms, risk factors, associated impairment, prognosis, and treatment options including behavioral interventions and medication.
  Arms: Training

SUMMARY:
The study aims to assess the impact of implementing ADHD knowledge improvement program on male primary school teachers' knowledge regarding ADHD in Abha City, Saudi Arabia.

DETAILED DESCRIPTION:
Primary school teachers play an essential role in early detection and proper treatment of school children suffering attention deficit hyperactivity disorder (ADHD). There are indications that teachers may not have enough knowledge about this disorder. Training programs can help to improve the knowledge of teachers about ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male teachers in governmental and private primary schools in Abha City, Saudi Arabia.

Exclusion Criteria:

* Those who have a similar training program before.
* Those who are not directly involved in the teaching process.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Teachers' Knowledge questionnaire | 1 month
  A self-administered questionnaire. The questionnaire composed of 6 items covering socio-demographic characteristics of teachers (age, nationality, years of experience, education level, specialty and type of school) and 20 items assessing teachers' knowledge of ADHD. Each item was assessed on a 2-point scale (incorrect response and don't know = 0, correct response = 1) with a maximum score of 20. The questionnaire items were as follows: nature of disease (1 item), age of onset (1 item), sex prevalence (1 item), disease course (1 item), symptoms (7 items), risk factors (4 items), aggravating factors (4 items) and management (1 item). Adequate knowledge was considered when the teachers achieved 65% of the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Abdullah Alshehri, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Polanczyk GV, Salum GA, Sugaya LS, Caye A, Rohde LA. Annual research review: A meta-analysis of the worldwide prevalence of mental disorders in children and adolescents. J Child Psychol Psychiatry. 2015 Mar;56(3):345-65. doi: 10.1111/jcpp.12381. Epub 2015 Feb 3. PMID 25649325
- [Background] Spencer TJ. ADHD and comorbidity in childhood. J Clin Psychiatry. 2006;67 Suppl 8:27-31. PMID 16961427
- [Background] Awadalla NJ, Ali OF, Elshaer S, Eissa M. Role of school teachers in identifying attention deficit hyperactivity disorder among primary school children in Mansoura, Egypt. East Mediterr Health J. 2016 Nov 2;22(8):586-595. doi: 10.26719/2016.22.8.586. PMID 27834440
- [Background] Moher D, Dulberg CS, Wells GA. Statistical power, sample size, and their reporting in randomized controlled trials. JAMA. 1994 Jul 13;272(2):122-4. PMID 8015121
- [Background] Muanprasart P, Traivaree C, Arunyanart W, Teeranate C. Knowledge of attention deficit hyperactivity disorder and its associated factors among teachers in 3 large primary schools in Phra Nakorn Sri Ayutthaya Province, Thailand. J Med Assoc Thai. 2014 Feb;97 Suppl 2:S107-14. PMID 25518183
- [Background] Alqahtani MM. Attention-deficit hyperactive disorder in school-aged children in Saudi Arabia. Eur J Pediatr. 2010 Sep;169(9):1113-7. doi: 10.1007/s00431-010-1190-y. Epub 2010 Mar 27. PMID 20339867
- [Background] Reebye P. Attention-Deficit Hyperactivity Disorder: A Handbook For Diagnosis And Treatment, Third Edition. J Can Acad Child Adolesc Psychiatry. 2008;17(1):31-33.
- [Background] Lasisi D, Ani C, Lasebikan V, Sheikh L, Omigbodun O. Effect of attention-deficit-hyperactivity-disorder training program on the knowledge and attitudes of primary school teachers in Kaduna, North West Nigeria. Child Adolesc Psychiatry Ment Health. 2017 Mar 20;11:15. doi: 10.1186/s13034-017-0153-8. eCollection 2017. PMID 28331540
- [Background] Sarraf N, Karahmadi M, Marasy MR, Azhar SM. A comparative study of the effectiveness of nonattendance and workshop education of primary school teachers on their knowledge, attitude and function towards ADHD students in Isfahan in 2010. J Res Med Sci. 2011 Sep;16(9):1196-201. PMID 22973389
- [Background] Homidi M, Obaidat Y, Hamaidi D. Prevalence of attention deficit and hyperactivity disorder among primary school students in Jeddah city, KSA. Life Sci J. 2013;10(3):280-5
- [Background] Alkahtani, K. (2013). Teachers' Knowledge and Misconceptions of Attention Deficit/Hyperactivity Disorder. Psychology, 4, 963-969. doi: 10.4236/psych.2013.412139.
- [Background] Al Hamed JH, Taha AZ, Sabra AA, Bella H. Attention Deficit Hyperactivity Disorder (ADHD) among Male Primary School Children in Dammam, Saudi Arabia: Prevalence and Associated Factors. J Egypt Public Health Assoc. 2008;83(3-4):165-82. PMID 19302773
- [Background] Ali Munshi AM. Knowledge and Misperceptions towards diagnosis and management of attention deficit hyperactivity disorder (ADHD) among Primary School and kindergarten female teachers in Al-Rusaifah district, Makkah city, Saudi Arabia. Int J Med Sci Public Health 2014;3:434-441.
- See also: Related Info — http://www.psychiatryonline.org